CLINICAL TRIAL: NCT03341832
Title: A Randomized, Double-blind, Active- and Placebo-controlled, Parallel, Multicenter, Phase II an Exploratory Clinical Trial to Evaluate the Efficacy and Safety NVP-1203 in Patients With Acute Low Back Pain
Brief Title: Efficacy and Safety of NVP-1203 in Patients With Acute Low Back Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NVP Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NVP-1203_P2
Record Dates: First submitted 2017-11-09; First posted 2017-11-14 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2018-02

CONDITIONS: Acute Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NVP-1203 (Experimental): NVP-1203 plus NVP-1203-R placebo for up to 7 days, oral dose
  Interventions: Drug: NVP-1203; Drug: NVP-1203-R placebo
- NVP-1203-R (Active Comparator): NVP-1203-R plus NVP-1203 placebo for up to 7 days, oral dose
  Interventions: Drug: NVP-1203-R; Drug: NVP-1203 placebo
- Placebo (Placebo Comparator): NVP-1203 placebo plus NVP-1203-R placebo for up to 7 days, oral dose
  Interventions: Drug: NVP-1203 placebo; Drug: NVP-1203-R placebo

INTERVENTIONS:
Drug: NVP-1203 — oral dose for 7 days
  Arms: NVP-1203
Drug: NVP-1203-R — oral dose for 7 days
  Arms: NVP-1203-R
Drug: NVP-1203 placebo — oral dose for 7 days
  Arms: NVP-1203-R; Placebo
Drug: NVP-1203-R placebo — oral dose for 7 days
  Arms: NVP-1203; Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety NVP-1203 in patients with Acute low back pain

DETAILED DESCRIPTION:
This study is a randomized, double-blind, active- and placebo-controlled, parallel, phase II study to evaluate efficacy and safety of NVP-1203 in patients with Acute low back pain

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have ability to comprehend the contents of study and before participating in trial and have willingness to sign of informed consent in writing
* 19 Years and older
* A patient has symptom of acute low back pain

Exclusion Criteria:

* Subjects who cannot prohibit anti-inflammatory drug or muscle relaxants during clinical trial
* Inadequate subject for the clinical trial by the investigator's decision

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2019-01-15 (Actual); Study Completion 2019-01-15 (Actual)

PRIMARY OUTCOMES:
VAS Pain Intensity | 3, 7 days
  Improvement in VAS compared to baseline

SECONDARY OUTCOMES:
Finger to Floor Distance (FFD) | 3, 7 days
  Improvement in FFD compared to baseline
Oswestry Disability Index(ODI) | 3, 7 days
  Improvement in ODI compared to baseline
Investigator Global Assessment of Response to Therapy(IGART) | 7 days
  Improvement in IGART compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Seong-Hwan Moon, MD, Principal Investigator — Severance Hospital; Jin Hwan Kim, MD, Principal Investigator — Inje University; Tae Kyun Kim, MD, Principal Investigator — Wonkwang University Hospital
Locations (1):
- Navipharm, Suwon, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No